CLINICAL TRIAL: NCT04374292
Title: Open Clinical Trial to Modify the Eating Habits of Children With Obesity, Comparing the Nutritional Family Intervention Versus the Usual Consultation
Brief Title: Dietary Habits and Metabolic Response in Obese Children Whose Mothers Received an Intervention to Promote Healthy Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Infantil de Mexico Federico Gomez (Other)
Responsible Party: Principal Investigator, Dr Salvador Villalpando-Carrion, Principal Investigator, Hospital Infantil de Mexico Federico Gomez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIM 2011-003
Record Dates: First submitted 2020-04-19; First posted 2020-05-05 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-03

CONDITIONS: Obesity; Child Obesity
Keywords: Feeding behavior; Intervention; Insulin resistance; Dietary habits; Childhood obesity
MeSH Terms: conditions — Obesity; Pediatric Obesity; Feeding Behavior; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: After providing written consent, 177 children with obesity (BMI ≥ 95 pc) of age 5-11 years and their mothers were randomly assigned to participate in the intervention group (IG) or the control group (CG). None of the participating children were receiving pharmacological treatment for obesity, were morbidly obese or were associated with a genetic syndrome. Intervention group mothers (n = 90) attended six weekly group sessions, which were led by nutritionists and lasted 90 minutes.
Masking Description: After providing written consent, 177 children with obesity (BMI ≥ 95 pc) of age 5-11 years and their mothers were randomly assigned to participate in the intervention group (IG) or the control group (CG).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group mothers (n = 90) attended six weekly group sessions, which were led by nutritionists and lasted 90 minutes.
  The key message was that healthy dietary habits and health risks are acquired at home and that opportunities for change can be identified in the processes that surround meal times. It begins with selecting and purchasing food, followed by preparation and consumption behaviors. Mothers were encouraged to participate in the sessions which involved the use of food models, videos, slides, and, in some cases, real food. Upon completing each session, mothers were given printed material to add to a home consultation manual.
  Upon concluding consultations and group sessions, mother/child pairs from both groups were asked to return for monthly follow-ups over the next three months.
  Interventions: Behavioral: Family intervention
- Control group (Active Comparator): Control group mothers and children (n = 87) were given the usual nutritional consultation and were prescribed diets that covered their energy requirements according to their age and sex. Similarly, CG mother/child pairs received information regarding food groups and portion sizes, were trained in the use of the food equivalence system to encourage variation, and were instructed on how to prepare the diet at home.
  Interventions: Other: Usual nutritional consultation

INTERVENTIONS:
Behavioral: Family intervention — Topics covered in each session with intervention group mothers.
  1. Dietary and physical activity habits and their link to obesity and cardio-metabolic diseases. Children learn about healthy eating habits and health risks at home.
  2. Food-preparation processes. Selecting and purchasing food and beverages; importance of food groups and their impact on health; importance of fruit and vegetables. Balance between food groups, source of foods, organic or industrialized. Family menu preparation.
  3. Habits and behaviors surrounding eating processes identified as health or risk factors, such as energy density, portion-size control, controlling emotional eating.
  4. Beverages. Water versus sugar-sweetened drinks prepared at home or purchased at the store.
  5. Preventing the risk of cardiovascular diseases by learning healthy eating habits and practicing these habits at home.
  6. Integration. Practicing the skills learned during the intervention in each stage of preparing food and eating
  Arms: Intervention group
Other: Usual nutritional consultation — Control group mothers and children (n = 87) were given the usual nutritional consultation and were prescribed diets that covered their energy requirements according to their age and sex. CG mother/child pairs received information regarding food groups and portion sizes, were trained in the use of the food equivalence system to encourage variation, and were instructed on how to prepare the diet at home.
  Arms: Control group

SUMMARY:
Unhealthy eating habits inside and outside the home lead to developing obesity, leading to clinical and metabolic disorders, such as insulin resistance, metabolic syndrome, and chronic degenerative diseases, which are the leading causes of death in adult life. The present study compared changes in dietary habits, behaviors and metabolic profiles of obese children whose mothers attended group sessions, with those who received the usual nutritional consultation.

The hypotheses were:

1. The mother's training in healthy eating methods, eliminating foods and nutrients that represent metabolic and cardiovascular risk, will change the consumption of these foods in the family, reducing them by 20% and increasing the consumption of food in the same proportion. beneficial, compared to the family of the child who only receives individual consultation.
2. Children with obesity who modify or eliminate metabolic and cardiovascular risk foods and nutrients from their normal diet will have a weight loss of -1.5 BMI compared to children who only receive the usual consultation.

Randomized clinical trial, 177 mother/obese child pairs participated, 90 in the intervention group (IG) and 87 in the control group (CG). The intervention group attended six group education sessions to promote healthy eating and 87 received the usual nutritional consultation, over a three-month period. Frequency of food consumption, behaviors during feeding in the house and metabolic profile was evaluated. Data was compared using Student's t or X2.

DETAILED DESCRIPTION:
The aim of this study is evaluate the change in eating behaviors, metabolic condition, and nutritional status measured by anthropometry, in children with obesity who were prescribed a diet to reduce their body weight in the usual nutritional consultation, in comparison to children whose mothers participated in an intervention of six group sessions to acquire healthy dietary habits.

Methods. Design. The Obesity Clinic at Federico Gómez Children's Hospital of Mexico conducted a randomized clinical trial between January 2011 and December 2014 with approval from the hospital's Research, Ethics and Biosecurity Committee. After providing written consent, 177 children with obesity (BMI ≥ 95 pc) of age 5-11 years and their mothers were randomly assigned to participate in the intervention group (IG) or the control group (CG). None of the participating children were receiving pharmacological treatment for obesity, were morbidly obese or were associated with a genetic syndrome. Intervention group mothers (n = 90) attended six weekly group sessions, which were led by nutritionists and lasted 90 minutes.

The key message was that healthy dietary habits and health risks are acquired at home and that opportunities for change can be identified in the processes that surround meal times. It begins with selecting and purchasing food, followed by preparation and consumption behaviors. Mothers were encouraged to participate in the sessions which involved the use of food models, videos, slides, and, in some cases, real food. Upon completing each session, mothers were given printed material to add to a home consultation manual. Children in this group were not prescribed diets to reduce their body weight. Control group mothers and children (n = 87) were given the usual nutritional consultation and were prescribed diets that covered their energy requirements according to their age and sex. Similarly, CG mother/child pairs received information regarding food groups and portion sizes, were trained in the use of the food equivalence system to encourage variation, and were instructed on how to prepare the diet at home. Neither group of children received physical activity programs. Upon concluding consultations and group sessions, mother/child pairs from both groups were asked to return for monthly follow-ups over the next three months.

The assignment to intervention or control groups was made using a block randomization with 8 mother/child pairs in each block to assure equal allocation to groups. One of coworkers not involved in data collection produced a computer-generated randomization list using the Stata 11.0 program. Children were randomized at the end of the baseline examination. Taking experiences from the published studies the sample size calculation was based on to expect differences of at less 20% in eating habits between the mothers/children dyad of the intervention or control groups, to detect differences with significant level of 5% and 80% power; the size of sample required was 72 mother/children pairs per group and to allow for 20% drop-out during the follow-up, the investigators aimed at recruiting 86 mother/children dyad per group.

Measurements at the beginning and end of the study. Anthropometry. The weight, height and waist circumference of children in both groups were measured according to international procedures. Weight was measured on a mechanical scale (Seca model-700, SECA Corp., Hamburg, Germany) with 50 g precision. Height was measured on a stadiometer (SECA model-225, SECA Corp., Hamburg, Germany) 0.1 cm precision. Meanwhile, waist circumference was measured at the end of an exhalation with non-elastic flexible tape (Seca model-200, SECA Corp., Hamburg, Germany) in a standing position at the midpoint between the lower costal border and the iliac crest. Body Mass Index (BMI) and percentile value were calculated using CDC data for reference, children with a BMI ≥ 95 pc were categorized with obesity.

Blood pressure. Blood pressure was measured on children's right arm with a mercury sphygmomanometer (ALPK2, Tokyo, Japan) using a cuff that suited arm length and perimeter and following 2004 National High Blood Pressure Education Program guidelines.

Questionnaires. A questionnaire of socio demographic data was applied to the mothers at baseline. In addition, a survey of family feeding habits at home at baseline and three months was applied, the mother was asked about the child's breakfast habit and bring lunch to consume at school, family feeding habits at the time of sitting at the table (place the salt shaker, sugar and sweetened soft drinks on the table, fill the plate, repeat saucer, force the child to finish the meal, accept the exchange of food to what the child wants), frequency of consumption of food (fried, roasted, fruits and vegetables) and drinks (simple water, sugary drinks prepared at home, natural juice, industrialized juice and soft drinks). The amounts of food consumption were not evaluated. A survey of physical activity and sedentary activities was applied; no physical activity intervention was performed during this study.

Blood sample. 5 mL venous blood samples after 12 h fasting periods were drawn to determine glucose (mg/dL)(hexokinase method Dimension RxL Max, Siemens Euro, DPC, Llanberis, UK), insulin (mIU/mL) (chemiluminescence IMMULITE 1000, Siemens), HDL cholesterol (mg/dl) (enzymatic reaction/catalase, using ADVIA ® 1800 equipment), and triglycerides (mg/dl) (ILAB 300, Instrumentation Laboratory, Barcelona Spain). Participating children's HOMA-IR index was obtained through glucose and insulin data (If xGf/22.5).

Statistical analysis. Central tendency measures were used to describe the study population's baseline characteristics. Student's t-test for independent samples was used to compare continuous variables, such as socio-demographic data, dietary habits, feeding behaviors, and biochemical and anthropometric data. Pearson X2 test was used to compare proportions between groups. Continuous data without normal distribution was managed using logarithmic transformation or square root. Student's t-test for related samples was used to identify differences before and after the intervention in each group or its non-parametric Wilcoxon equivalent. The equal proportions test was used to assess the difference in proportions in dietary habits and behaviors between groups. Statistical significance was considered at P < 0.05. Analyses were carried out with STATA SE v.12.0 (Stata Corp, CollegeStation, TX, USA).

ELIGIBILITY:
Inclusion Criteria:

* Children and their families who come to the obesity clinic of the Federico Gómez Children's Hospital in Mexico who live in Mexico City or in the metropolitan area.
* Aged 5 to 11 years, both sexes.
* Children who can attend a consultation on a monthly basis for 3 months.
* Children and parents who have given their informed consent and assent in writing.

Exclusion Criteria:

* Children with obesity who receive medications that alter their body composition such as steroids, antiretrovirals and appetite stimulants.
* Children who are already under nutritional, medical or pharmacological treatment for their obesity.
* Children with syndromes whose body composition is altered, such as Cushing and other genetics.

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2011-01-05 (Actual); Primary Completion 2013-07-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in HOMA-IR | It was determined at the beginning of the study and at the end of the intervention (0 and 3 months)
  Change in Homeostasis Model to Assess the Insulin Resistance Index
Relative percentage obtained from the change in eating habits at the start of the study at 3 months. | It was measure at baseline and three months
  Changes in eating habits at home were obtained using the relative percentage. The change was obtained by comparing the initial percentage of each habit (100%) (baseline) versus the final percentage of the eating habit (3 months).
  Feeding habits are:
  * Breakfast
  * Habits at lunchtime: Putting salt on the table, putting sugar on the table, putting sweet soft drinks on the table, serves the right portion filling the food plate, repeating portion, forcing to finish food, accepting food substitutions,
  * Frequency of food consumption: fried foods (> 3times/wk), roasted foods, fruits, vegetables, frequency of beverage, simple water, sweetened water prepared at home, natural juice, industrialized juice, soft drinks
  * Time to finish food
  * Children watching TV at mealtime

SECONDARY OUTCOMES:
Change in BMI percentile | It was measure at baseline and three months
  Change in Body mass index percentile

CONTACTS AND LOCATIONS:
Overall Officials: Iris Nayeli López-Contreras, MSc, Principal Investigator — Hospital Infantil de Mexico Federico Gomez

IPD SHARING:
Plan to Share IPD: Yes
The results obtained from the study will be analyzed and published in an international indexed journal.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The results of the study will be published in an international indexed journal, approximately in July 2020.
Access Criteria: The results will be available to the public and the scientific community from the publication of the article.

REFERENCES:
- [Background] Vilchis-Gil J, Klunder-Klunder M, Duque X, Flores-Huerta S. Decreased Body Mass Index in Schoolchildren After Yearlong Information Sessions With Parents Reinforced With Web and Mobile Phone Resources: Community Trial. J Med Internet Res. 2016 Jun 24;18(6):e174. doi: 10.2196/jmir.5584. PMID 27342650
- [Derived] Lopez-Contreras IN, Vilchis-Gil J, Klunder-Klunder M, Villalpando-Carrion S, Flores-Huerta S. Dietary habits and metabolic response improve in obese children whose mothers received an intervention to promote healthy eating: randomized clinical trial. BMC Public Health. 2020 Aug 14;20(1):1240. doi: 10.1186/s12889-020-09339-4. PMID 32795294
- See also: PDF of paper — http://www.jmir.org/2016/6/e174/pdf